CLINICAL TRIAL: NCT03966430
Title: Jinling Hospital, Medical School of Nanjing University
Brief Title: Damage Control Surgery in Acute Mesenteric Ischemia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gao Tao (Other)
Responsible Party: Sponsor-Investigator, Gao Tao, Clinical Professor, Nanjing PLA General Hospital
Organization: Nanjing PLA General Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014NZGKJ-020
Record Dates: First submitted 2019-05-14; First posted 2019-05-29 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Damage Control
Keywords: damage control surgery; acute mesenteric ischemia; complication

STUDY DESIGN:
Intervention Model Description: a single center prospective cohort study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- damage control surgery group (Experimental): According to the discussion between the patient and the doctor, the patient signed the consent form and voluntarily enrolled and subsequently the patient was included in the damage control surgery group.
  Interventions: Procedure: damage control surgery
- non-damage control surgery group (Sham Comparator): According to the discussion between the patient and the doctor, the patient signed the consent form and voluntarily enrolled and subsequently the patient was included in the non-damage control surgery group.
  Interventions: Procedure: non-damage control surgery

INTERVENTIONS:
Procedure: damage control surgery — 1. Emergency surgery stage, (a) the hybrid operating room restores mesenteric vascular patency. (b) excision of the necrotic intestine (c) retention of suspicious intestinal ducts, double stoma (d) establishment of catheter thrombolysis pathway (e) apply TAC to maintain open abdominal.
  2. ICU phase, including (a) fluid resuscitation; (b) anti-infective and organ function support therapy; (c) continued local anticoagulation, thrombolysis (d) arrange planned re-laparotomy (e) early EN.
  3. Definitive surgical procedures, including (a) Deterministic fascia closure or further removal of the necrotic intestine. (b) Intestinal stoma care and enteral nutrition support treatment. (c) An enterostomy was performed about 6 months after the first operation.
  Arms: damage control surgery group
Procedure: non-damage control surgery — The patients are diagnosed with AMI and treated for mesenteric thrombosis and ischemic bowel.
  1. The patient retains the endoluminal catheter after the DSA was diagnosed as AMI.
  2. After diagnosis, the operation is performed in the general operating room, and the intestinal fistula double or the anastomosis is performed according to the judgment of the surgeon.
  3. After the operation, re-laparotomy is performed on demand.
  Arms: non-damage control surgery group

SUMMARY:
Acute mesenteric ischemia (AMI) is a rare but catastrophic abdominal vascular emergency associated with daunting mortality comparable to myocardial infarction or cerebral stroke. Damage control surgery has been extensively used in severe traumatic patients. Very urgent, there was no large-scale in-depth study when extended to a nontrauma setting, especially in the intestinal stroke center. Recently, the liberal use of OA as a damage control surgery adjunct has been proved to improve the clinical outcome in acute superior mesenteric artery occlusion patients. However, there was little information when extended to a prospective study. The purpose of this prospective cohort study was to evaluate whether the application of damage control surgery concept in AMI was related to avoiding postoperative abdominal infection, reduced secondary laparotomy, reduced mortality and improved the clinical outcomes in short bowel syndrome.

DETAILED DESCRIPTION:
Acute mesenteric ischemia (AMI) is a rare but catastrophic abdominal vascular emergency associated with daunting mortality comparable to myocardial infarction or cerebral stroke. Computed tomographic angiography is the initial diagnostic examination of choice for patients in whom AMI is a consideration. Computed tomographic angiography can be performed rapidly and can be used to identify critical arterial stenosis or occlusion as well as providing information concerning the presence of bowel infarction. An uncommon cause of presentation to emergency rooms, lack of clinical suspicion often leads to delayed presentation, development of peritoneal signs, and subsequent staggeringly high mortality rates.

Now in use for over 2 decades, the concept of damage control surgery (DCS) has become an accepted, proven surgical strategy with wide applicability and success in severe trauma patients. The concept has been mostly used in the massively injured, exsanguinating patients with multiple competing surgical priorities. With growing experiences in the application, the strategy continues to evolve into a nontrauma setting, especially in AMI.

Although an increasing development of endovascular techniques, AMI remains a morbid condition with a poor short-term and long-term survival rate. Some authors advocated that laparotomy after mesenteric revascularization serves to evaluate the possible damage to the visceral organs. Bowel resection as a result of transmural necrosis is carried out according to the principles of DCS. Bowel resections are performed with staples, leaving the creation of stomas until the second-look laparotomy. The abdominal wall can be left unsutured and temporary abdominal closure (TAC) was applied. However, the use of DCS in the setting of AMI was limited in case series and mostly confined in large university teaching hospitals. The timing and details of how the DCS incorporated into the treatment algorithm of AMI deserved further investigations.

An integrated intestinal stroke center (ISC) was established in our department, a national cutting-edge referral center for intestinal failure, to build up ideal coordination among gastroenterology physician, gastrointestinal and vascular surgeon, and intervention radiologist for this therapeutic challenge. DCS was liberally used since ISC was established in 2010.

In this prospective cohort study, we aimed to compare the clinical outcomes of patients receiving DCS and non-DCS in the devastating conditions in our single center.

ELIGIBILITY:
Inclusion Criteria:

* Subjects and their families voluntarily and sign the informed consent form for this trial;
* Age is greater than or equal to 18 years old, less than or equal to 75 years old;
* Patients diagnosed with AMI;
* Subjects can objectively describe the symptoms and follow the follow-up plan.

Exclusion Criteria:

* Those who are judged by the physician to be unfit to participate in the test;
* non-obstructive mesenteric ischemia;
* Aortic dissection complicated with visceral ischemia;
* Intestinal ischemia secondary to other causes (such as volvulus, intestinal adhesion, strangulation);
* There is irreversible heart failure, liver failure or renal failure before diagnosis;
* History of intestinal ischemia surgery or complex abdominal surgery;
* Patients who are unable to perform surgical treatment for injury control or have surgical contraindications for significant injury control;
* Pregnancy, lactating women, subjects with a pregnancy plan within 1 month after the test (including male subjects);
* Participate in other clinical trials within 3 months before the trial;
* Transfer to the hospital within 1 week or discharge automatically;
* Sponsors or researchers or their family members who are directly involved in the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-01-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative 30-day mortality | 30 days
  All cause mortality within 30 days
Rate of postoperative abdominal sepsis | 30 days
  All cause postoperative abdominal infection
Rate of postoperative re-laparotomy | 30 days
  All cause postoperative re-laparotomy
Postoperative short bowel syndrome rate | 30 days
  All cause postoperative short bowel syndrome

SECONDARY OUTCOMES:
Rate of abdominal septic complications | 30 days
  Including wound infections, anastomotic leakage/anastomotic fistula, and intra-abdominal abscess
Rate of non-abdominal septic complications | 30 days
  Including thromboembolic complications
Rate of abdominal non-septic complications | 30 days
  including pneumonia and urinary tract infections
Rate of systematic complications | 30 days
  including thromboembolic complications
Length of preoperative stay | 30 days
  Number of days from admission to operation
Operative information | 30 days
  Including postoperative diagnosis, surgical name, surgical procedure (laparoscopic, open)
Recovery of intestinal function | 30 days
  first ventilation time after surgery (length in days), first defecation time (length in days), first recovery of semi-flow diet time (length in days);
The amount of nutritional support treatment | 30 days
  The amount (ml) of nutritional support daily
Catheter condition | 30 days
  whether to indwell the stomach tube (yes, no) with its extraction time (day)
Postoperative activity time | 30 days
  Time (hour) of getting out of bed every day after surgery;
Inflammatory markers | Postoperative day-1, 3, 5, 7
  Serum IL-6 and CRP levels in preoperative and postoperative patients
Infectious markers | Postoperative day-1, 3, 5, 7
  Pre- and post-operative patients with procalcitonin levels
Coagulation markers | Postoperative day-1, 3, 5, 7
  Blood PT, APTT, INR levels before and after surgery
Fibrinolytic markers | Postoperative day-1, 3, 5, 7
  Blood D-dimer, FDP levels before and after surgery
Intestinal barrier function markers | Postoperative day-1, 3, 5, 7
  Urinary citrulline and I-FABP in preoperative and postoperative patients
General nutritional information measurement | Postoperative day-1, 3, 5, 7
  Preoperative and postoperative patient weight (kg) and weight change (kg);
Immunological markers | Preoperative day-1 and postoperative day-1, 3, 5, 7
  Levels of blood T cell subsets (including CD3+ (%), CD4+ (%), and CD4+/CD8+);
Re-admission rate 30 days after discharge | 30 days
  Re-admission time (day), cause;
Postoperative hospital stay | 1 year
  Number of days in hospital (day)
Postoperative ICU stay | 1 year
  Number of days in ICU (day)
Hospital costs | 1 year
  Cost from the hospital's financial system statistics (RMB)
Intraoperative intestinal length | 30 days
  length of intestine (length in centimetre), length of remaining intestine (length in centimetre)
Type of intestinal anastomosis | 30 days
  whether one-stage anastomosis (yes, no)
Operation time | 30 days
  operation time (hour)
Amount of fluid input and output during operation | 30 days
  intraoperative blood loss (ml), surgery Middle infusion volume (ml), intraoperative blood transfusion volume (ml)
Embolus size measurement | 30 days
  embolus size (cm)
Type of abdominal closure | 30 days
  (normal, temporary abdominal closure)
Type of abdominal drainage | 30 days
  abdominal drainage tube (yes, no) with an extraction time (day)
The time of nutritional support treatment | 30 days
  The start and end time of parenteral nutrition and enteral nutrition (days);
Degree of postoperative activity | 30 days
  Distance (m) of getting out of bed every day after surgery;
Serum nutrition marker | Postoperative day-1, 3, 5, 7
  Preoperative and postoperative serum albumin (g/L), prealbumin (mg/L), transferrin (g/L), hemoglobin (g/L), white blood cell count (10^9/L), platelet count (10^9/L), and hematocrit (L/L);
Marker of neutrophil extracellular traps markers | Preoperative day-1 and postoperative day-1, 3, 5, 7
  Levels of blood neutrophil extracellular traps markers (including CitH3 (IU/mL), cf-DNA (ng/mL), MPO-DNA (Abs405)) levels
The composition of nutritional support treatment | 30 days
  Composition of enteral nutrition daily (%)

CONTACTS AND LOCATIONS:
Locations (1):
- Jinling Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
IPD can be shared with the consent of the hospital patient information management department and the clinical trial leader.